CLINICAL TRIAL: NCT01619605
Title: The Utility of Serum Tryptase in the Diagnosis of Shrimp- Induced Anaphylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 669/2551(EC4)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Food (Shrimp) Allergy
Keywords: tryptases; anaphylaxis; shrimp allergy
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shrim (Experimental)
  Interventions: Procedure: shrimp challenge

INTERVENTIONS:
Procedure: shrimp challenge — Patients with history of shrimp allergy and positive skin tests to shrimp were recruited for shrimp challenges After shrimp challenges, patients with anaphylaxis defined as anaphylaxis group, patients with mild reactions defined as mild reaction group, and patients without symptom defined as control group
  Other Names: open food challenge

SUMMARY:
The purpose of this study was to investigate the utility of serum tryptase for the confirmation of shrimp-induced anaphylaxis.

DETAILED DESCRIPTION:
The diagnosis of anaphylaxis is based primarily on the clinical history. In some circumstances, inability to confirm the clinical diagnosis such as present with unusual manifestation, or when skin signs are absent likely contributes to underrecognition and undertreatment of the disease.

Currently, products of mast cell activation (histamine and total tryptase) can be measure in clinical laboratories as markers of acute anaphylaxis events, however these tests have clinically relevant limitations.

Therefore, development of laboratory tests with improved sensitivity and specificity that will support the clinical diagnosis of anaphylaxis are needed.

In addition, shrimp is the major cause of seafood anaphylaxis among Thai children.

ELIGIBILITY:
Inclusion Criteria:

* a history of shrimp allergy

Exclusion Criteria:

* severe anaphylactic reaction from seafood
* pregnancy
* underlying diseases such as cardiovascular, hepatobiliary, and renal diseases
* on systemic corticosteroid or β-blocking agents

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change of Serum tryptases | baseline and 60 minutes after the onset of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Orathai Piboonpocanun, Assoc.Prof., Principal Investigator — Mahidol University
Locations (1):
- Pediatric allergy clinic, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand